CLINICAL TRIAL: NCT00189670
Title: A Phase II Randomized Trial of 6 TEC Every 3 Weeks, Versus 4 EC Followed by 4 Taxotere Every 2 Weeks, Versus 4 Taxotere Followed by 4 EC Every 2 Weeks in Node Positive Breast Cancer
Brief Title: Randomized Phase II Trial of Dose Dense Docetaxel in N+ Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Association Européenne de Recherche en Oncologie (Other)
Collaborators: Aventis Pharmaceuticals (Industry); Amgen (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AERO-B03
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2005-09-19 (Estimated); Status verified 2005-09

CONDITIONS: Node Positive Breast Cancer

INTERVENTIONS:
Procedure: 6 TEC q 3 weeks
Procedure: 4 EC q 2 weeks followed by 4 TXT q 2 weeks
Procedure: 4 TXT q 2 weeks followed by 4 EC q 2 weeks

SUMMARY:
To screen a dose-dense arm to be used in a future large scale phase III trial. Primary endpoint is safety; secondary endpoints are disease free survival and overall survival. A total of 100 patients were included.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically proven breast cancer
* Surgical resection performed with clear margins (R0 resection)
* At least 1 histologically proven involved axillary node
* ER + or ER-
* Interval between surgery (2nd surgical procedure in case of multiple procedures) and randomization inferior to 60 days
* Aged over 18 years, and more than 10-year life expectancy
* ECOG performance status 0-1
* Signed informed consent form prior to randomization

Exclusion Criteria:

* Bilateral breast cancer
* Inflammatory breast cancer
* Personal history of breast cancer
* Immunohistochemical only node involvement
* Intraductal breast cancer
* Distant metastases
* Contraindication to any drug contained in the chemotherapy regimens
* Any serious active disease or co-morbid medical condition including recent history of severe sepsis and digestive inflammatory disease
* Poor renal function (creatinin level > 120 micromol/L), poor hepatic function (total bilirubin level > 1 UNL), transaminases > 2.5 UNL)
* Poor bone marrow reserve as defined by neutrophils < 1.5 G/L or platelets < 100 G/L; Hemoglobin < 10 G/dL
* Poor contractile cardiac function (LVEF < 50%)
* Coronary disease
* Any history of cancer during the last 5 years, with the exception of basal cell carcinomas or stage 0 (in situ) cervical carcinoma
* Pregnancy or breast feeding
* Absence of contraception in non menopausal women
* Adult patient unable to give informed consent because of intellectual impairment
* Concomitant participation to another trial

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Piedbois, MD, PhD, Principal Investigator — Association Europeenne de Recherche en Oncologie